CLINICAL TRIAL: NCT03574623
Title: Contralaterally Controlled FES Versus Cyclic NMES for Hand Function After Stroke
Brief Title: Therapies for Recovery of Hand Function After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Kessler Foundation (Other); National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); The Cleveland Clinic (Other); Johns Hopkins University (Other); Emory University (Other)
Responsible Party: Principal Investigator, Jayme Knutson, Senior Staff Scientist, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB17-00884; R01HD092351 (NIH)
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Upper Extremity Paresis; Hemiplegia
Keywords: stroke; rehabilitation; therapy; electrical stimulation; hand
MeSH Terms: conditions — Stroke; Paresis; Hemiplegia | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CCFES (Experimental): Contralaterally Controlled Functional Electrical Stimulation (CCFES) uses an electrical stimulator and surface electrodes placed over the paretic finger and thumb extensors to deliver stimulation with an intensity that is proportional to the degree of opening of the contralateral unimpaired hand wearing an instrumented glove. Thus, volitional opening of the nonparetic hand produces stimulated opening of the paretic hand. During the lab visits, participants in the CCFES group will use CCFES to assist hand opening during occupational therapy task practice. During their home sessions, participants in the CCFES group will use CCFES to perform hand opening exercise.
  Interventions: Device: Electrical Stimulator; Behavioral: Occupational Therapy
- cNMES (Active Comparator): Cyclic Neuromuscular Electrical Stimulation (cNMES) uses an electrical stimulator and surface electrodes over the paretic finger and thumb extensors to deliver electrical stimulation to open the weak hand. The stimulation automatically turns on and off causing the weak hand to open repetitively for several seconds at a time. During the lab visits, participants in the cNMES group will receive occupational therapy task practice. During their home sessions, participants in the cNMES group will use cNMES to perform hand opening exercise.
  Interventions: Device: Electrical Stimulator; Behavioral: Occupational Therapy
- Task Oriented Therapy (Active Comparator): Task Oriented Therapy (TOT) focuses on practicing using the weak hand to practice activities of daily living tasks. During the clinic visits, participants in the TOT group will receive occupational therapy task practice. During their home sessions, participants in the TOT group will practice using their hand to complete a list of tasks given to them by the therapist to ensure that the participant receives a high dose of task practice.
  Interventions: Behavioral: Occupational Therapy

INTERVENTIONS:
Device: Electrical Stimulator — An electrical stimulator will be used to deliver electrical current through surface electrodes to produce hand opening by making the paretic finger and thumb extensor muscles contract. The stimulator can be programmed to turn on and off in a repetitive cyclic fashion (i.e., cNMES) or be programmed to deliver stimulation with an intensity that corresponds to the opening of a glove instrumented with sensors and plugged into the stimulator (i.e., CCFES).
  Arms: CCFES; cNMES
Behavioral: Occupational Therapy — Task practice that requires movement and use of the paretic hand under the guidance of a trained therapist.

SUMMARY:
After a stroke, it is very common to lose the ability to open the affected hand. The purpose of this study is to compare the effects of three different therapies on recovery of hand function after stroke and determine if any one is better than the other.

DETAILED DESCRIPTION:
A single-blinded randomized controlled trial will be carried out to assess and compare the effects of 12 weeks of Contralaterally Controlled Functional Electrical Stimulation (CCFES), Cyclic Neuromuscular Electrical Stimulation (cNMES), and Task Oriented Training. Dexterity, upper limb impairment, and activity limitation will be assessed at 0 (baseline), 12 (end of treatment), and 36 weeks. The treatment dose will be the same for all three groups: 10 sessions per week of self-administered treatment at home plus 2 sessions per week of group-specific occupational therapy in the lab.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 24 months since a first clinical cortical or subcortical, hemorrhagic or nonhemorrhagic stroke
* unilateral upper limb hemiparesis with finger extensor strength of grade no more than 4 out of 5 on the Medical Research Council (MRC) scale
* score of at least 1 and no more than 11 out of 14 on the hand section of the upper extremity Fugl-Meyer Assessment
* adequate active movement of the shoulder and elbow to position the hand in the workspace for table-top task practice (necessary for the lab task practice sessions)
* able to follow 3-stage commands
* able to recall at least 2 of a list of 3 items after 30 minutes
* skin intact on the hemiparetic arm
* surface stimulation of the paretic finger and thumb extensors produces functional hand opening without pain (this will exclude those who have too much flexor spasticity)
* able to hear and respond to cues from stimulator
* not receiving occupational therapy (no concomitant OT)
* full voluntary opening/closing of the contralateral (less affected) hand
* demonstrates ability to follow instructions for operating the stimulator or have a caregiver who will assist them

Exclusion Criteria:

* co-existing neurologic diagnosis of peripheral nerve injury, Parkinson's disease, spinal cord injury, traumatic brain injury, or multiple sclerosis
* uncontrolled seizure disorder
* brainstem stroke
* uncompensated hemineglect
* severe shoulder or hand pain
* insensate forearm or hand
* history of potentially fatal cardiac arrhythmias with hemodynamic instability
* implanted electronic systems (e.g. pacemaker)
* botulinum toxin injections to any upper extremity muscle within 3 months of enrolling
* pregnant women due to unknown risks of surface NMES during pregnancy
* lack of functional passive range of motion of the wrist or fingers of affected side
* diagnosis (apart from stroke) that substantially affects paretic arm and hand function
* deficits in communication that interfere with reasonable study participation
* lacking sufficient visual acuity to see the stimulator's display
* concurrent enrollment in another investigational study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Box and Blocks Test (BBT) change | 0 to 12 weeks, 0 to 36 weeks
  The BBT is a measure of hand dexterity. It is a count of how many blocks a patient can pick up, move over a barrier, and release in 60 seconds. The higher the score, the better the motor recovery.

SECONDARY OUTCOMES:
Upper Extremity Fugl Meyer (UEFM) change | 0 to 12 weeks, 0 to 36 weeks
  The UEFM is a measure of upper limb motor impairment with a maximum score of 66. The higher the score, the better the motor recovery.
Action Research Arm Test (ARAT) change | 0 to 12 weeks, 0 to 36 weeks
  The ARAT is a measure of arm and hand function with a maximum score of 57. The higher the score, the better the motor recovery.
Stroke Upper Limb Capacity Scale (SULCS) change | 0 to 12 weeks, 0 to 36 weeks
  The SULCS is a measure of upper limb capacity with a maximum score of 10. The higher the score, the better the motor recovery.
Responder Rate | 0 to 36 weeks
  Proportion of participants who had a gain of at least 6 points on the UEFM

CONTACTS AND LOCATIONS:
Overall Officials: Jayme Knutson, PhD, Principal Investigator — MetroHealth Medical Center
Locations (4):
- United States (4):
  - Emory University and Atlanta VA, Atlanta, Georgia
  - Johns Hopkins University, Baltimore, Maryland
  - Kessler Foundation, West Orange, New Jersey
  - MetroHealth Rehabilitation Institute, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knutson JS, Friedl AS, Hansen KM, Harley MY, Hogan SD, Cunningham DA, Hisel TZ, Plow EB, Barrett AM, Raghavan P, Boukrina O, Nahab F, Gunzler DD, Chae J. Contralaterally Controlled Functional Electrical Stimulation for Upper Extremity Recovery Following Stroke: A Multisite Randomized Controlled Trial. Stroke. 2025 Nov 13:10.1161/STROKEAHA.125.052891. doi: 10.1161/STROKEAHA.125.052891. Online ahead of print. PMID 41230603
- [Derived] Knutson JS, Friedl AS, Hansen KM, Harley MY, Barrett AM, Raghavan P, Plow EB, Gunzler DD, Chae J. Efficacy of contralaterally controlled functional electrical stimulation compared to cyclic neuromuscular electrical stimulation and task-oriented training for recovery of hand function after stroke: study protocol for a multi-site randomized controlled trial. Trials. 2022 May 12;23(1):397. doi: 10.1186/s13063-022-06303-y. PMID 35549747